CLINICAL TRIAL: NCT03920254
Title: A 3-Year, Multi-Center, Long-Term Safety (LTS) Study to Evaluate the Safety and Tolerability of TD-1473 in Subjects With Ulcerative Colitis (UC)
Brief Title: TD-1473 Long-Term Safety (LTS) Ulcerative Colitis (UC) Study
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Stopped early due to company decision. Company decision based on interim analysis results in TD-1473-0157.
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0164; 2018-002135-19 (EudraCT Number)
Record Dates: First submitted 2019-03-28; First posted 2019-04-18 (Actual); Results first posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Ulcerative Colitis (UC)
Keywords: TD-1473; Janus kinase inhibitor; JAK inhibitor; Inflammatory Bowel Disease; IBD; Ulcerative colitis; UC; Intestinal restriction; Gut-selective
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Long Term Safety (LTS)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Active Treatment TD-1473 with Dose A (Experimental): Oral daily dose of TD-1473 for up to 156 weeks
  Interventions: Drug: TD-1473 Dose A
- Active Treatment TD-1473 with Dose B (Experimental): Oral daily dose of TD-1473 for up to 156 weeks
  Interventions: Drug: TD-1473 Dose B
- Active Treatment TD-1473 with Dose C (Experimental): Oral daily dose of TD-1473 for up to 156 weeks
  Interventions: Drug: TD-1473 Dose C

INTERVENTIONS:
Drug: TD-1473 Dose A — See Arm description
  Arms: Active Treatment TD-1473 with Dose A
Drug: TD-1473 Dose B — See Arm description
  Arms: Active Treatment TD-1473 with Dose B
Drug: TD-1473 Dose C — See Arm description
  Arms: Active Treatment TD-1473 with Dose C

SUMMARY:
A 3-Year Multi-Center, Long-Term Safety (LTS) Study to Evaluate the Safety and Tolerability of TD-1473 in Subjects with Ulcerative Colitis who have participated in the Maintenance Study of Protocol 0157

DETAILED DESCRIPTION:
This is a multi-center, long-term safety study to evaluate the safety and tolerability of TD-1473 for up to 156 weeks (3 years) + 4 week follow-up in subjects with moderate to severe UC exiting the preceding Maintenance Study of Protocol 0157 (NCT03758443).

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, subjects are required to enter the LTS Study within 14 days of exiting the Maintenance Study of Protocol 0157 and must meet all the following criteria:

* Capable of providing informed consent, which must be obtained prior to any study related procedures.
* One of the following:

  * Those who demonstrated persistent loss of response (no improvement 8 weeks after meeting loss of response criteria) OR
  * Two Clinical Flares after an episode of loss of response during the Maintenance Study OR
  * Those who have completed the Maintenance Study and confirmation of clinical remission status results are available
* During the study and for 7 days after receiving the last dose of the study drug, females of childbearing potential or men capable of fathering children must agree to use highly effective birth control measures (failure rate <1% when used consistently and correctly)) or agree to abstain from sexual intercourse. Females of childbearing potential must test negative for pregnancy at Day 1
* All male subjects must agree to refrain from semen donation during the study and for 7 days after the last dose of study drug.
* Must be able and willing to adhere to the study visit schedule and comply with other study requirements.

Exclusion Criteria:

* Has symptoms suggestive of fulminant colitis, megacolon or intestinal perforation
* Likely to require surgery for UC or other major surgeries
* Has previously received / is currently receiving prohibited medications
* Has been diagnosed during Protocol 0157 with Crohn's disease, other colitis conditions or the subject has a current or past diagnosis of a fistula or abdominal abscess
* Has endoscopic findings during Protocol 0157 of colitis-associated colonic dysplasia (with the exception of subjects with non-colitis associated spontaneous adenomas that have been completely resected)
* Has clinically significant abnormalities in laboratory evaluations
* Additional exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 46 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Theravance Biopharma
Locations (160):
- United States (35):
  - Theravance Biopharma Investigational Site, Chula Vista, California
  - Theravance Biopharma Investigational Site, Lancaster, California
  - Theravance Biopharma Investigational Site, Orange, California
  - Theravance Biopharma Investigational Site, Colorado Springs, Colorado
  - Theravance Biopharma Investigational Site, Aventura, Florida
  - Theravance Biopharma Investigational Site, Clearwater, Florida
  - Theravance Biopharma Investigational Site, Largo, Florida
  - Theravance Biopharma Investigational Site, Miami, Florida
  - Theravance Biopharma Investigational Site, New Port Richey, Florida
  - Theravance Biopharma Investigational Site, New Smyrna Beach, Florida
  - Theravance Biopharma Investigational Site, Orlando, Florida
  - Theravance Biopharma Investigational Site, Pembroke Pines, Florida
  - Theravance Biopharma Investigational Site, Atlanta, Georgia
  - Theravance Biopharma Investigational Site, Suwanee, Georgia
  - Theravance Biopharma Investigational Site, Idaho Falls, Idaho
  - Theravance Biopharma Investigational Site, Kansas City, Kansas
  - Theravance Biopharma Investigational Site, Louisville, Kentucky
  - Theravance Biopharma Investigational Site, Monroe, Louisiana
  - Theravance Biopharma Investigational Site, Baltimore, Maryland
  - Theravance Biopharma Investigational Site, Troy, Michigan
  - Theravance Biopharma Investigational Site, Wyoming, Michigan
  - Theravance Biopharma Investigational Site, Rochester, Minnesota
  - Theravance Biopharma Investigational Site, Kansas City, Missouri
  - Theravance Biopharma Investigational Site, Las Vegas, Nevada
  - Theravance Biopharma Investigational Site, Charlotte, North Carolina
  - Theravance Biopharma Investigational Site, Gastonia, North Carolina
  - Theravance Biopharma Investigational Site, Greenville, North Carolina
  - Theravance Biopharma Investigational Site, Pittsburgh, Pennsylvania
  - Theravance Biopharma Investigational Site, Smithfield, Pennsylvania
  - Theravance Biopharma Investigational Site, Greenville, South Carolina
  - Theravance Biopharma Investigational Site, Rock Hill, South Carolina
  - Theravance Biopharma Investigational Site, Nashville, Tennessee
  - Theravance Biopharma Investigational Site, Garland, Texas
  - Theravance Biopharma Investigational Site, Houston, Texas
  - Theravance Biopharma Investigational Site, San Antonio, Texas
- Australia (4):
  - Theravance Biopharma Investigational Site, South Brisbane, Queensland
  - Theravance Biopharma Investigational Site, Woolloongabba, Queensland
  - Theravance Biopharma Investigational Site, Malvern, Victoria
  - Theravance Biopharma Investigational Site, Murdoch, Western Australia
- Bulgaria (9):
  - Theravance Biopharma Investigational Site, Sofia, Sofia
  - Theravance Biopharma Investigational Site #2, Pleven
  - Theravance Biopharma Investigational Site, Pleven
  - Theravance Biopharma Investigational Site, Plovdiv
  - Theravance Biopharma Investigational Site, Rousse
  - Theravance Biopharma Investigational Site, Sliven
  - Theravance Biopharma Investigational Site, Sofia
  - Theravance Biopharma Investigational Site, Stara Zagora
  - Theravance Biopharma Investigational Site, Veliko Tarnovo
- Theravance Biopharma Investigational Site, Kingston, Ontario, Canada
- France (9):
  - Theravance Biopharma Investigational Site, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Theravance Biopharma Investigational Site, Saint-Etienne, Auvergne-Rhône-Alpes
  - Theravance Biopharma Investigational Site, Reims, Champagne-ardenne
  - Theravance Biopharma Investigational Site, Lille, Hauts-de-France
  - Theravance Biopharma Investigational Site, Montpellier, Languedoc-roussillon
  - Theravance Biopharma Investigational Site, Vandœuvre-lès-Nancy, Limousin
  - Theravance Biopharma Investigational Site, Toulouse, Midi-pyrenees
  - Theravance Biopharma Investigational Site, Nantes, Pays de la Loire Region
  - Theravance Biopharma Investigational Site, Amiens, Picardie
- Georgia (2):
  - Theravance Biopharma Investigational Site, Batumi
  - Theravance Biopharma Investigational Site, Tbilisi
- Germany (3):
  - Theravance Biopharma Investigational Site, Heidelberg, Baden-Wurttemberg
  - Theravance Biopharma Investigational Site, Kiel, Schleswig-Holstein
  - Theravance Biopharma Investigational Site, Berlin
- Greece (4):
  - Theravance Biopharma Investigational Site, Athens, Attica
  - Theravance Biopharma Investigational Site #2, Athens, Attica
  - Theravance Biopharma Investigational Site, Heraklion, Crete
  - Theravance Biopharma Investigational Site, Patra, Peloponnese
- Hungary (4):
  - Theravance Biopharma Investigational Site, Székesfehérvár, Fejér
  - Theravance Biopharma Investigational Site, Debrecen, Hajdú-Bihar
  - Theravance Biopharma Investigational Site, Szekszárd, Tolna County
  - Theravance Biopharma Investigational Site, Budapest
- Israel (7):
  - Theravance Biopharma Investigational Site, Ẕerifin, Rehoboth
  - Theravance Biopharma Investigational Site, Haifa
  - Theravance Biopharma Investigational Site, Holon
  - Theravance Biopharma Investigational Site, Jerusalem
  - Theravance Biopharma Investigational Site, Nahariya
  - Theravance Biopharma Investigational Site, Petah Tikva
  - Theravance Biopharma Investigational Site, Rehovot
- Italy (3):
  - Theravance Biopharma Investigational Site, Rozzano, Milano
  - Theravance Biopharma Investigational Site, Catanzaro
  - Theravance Biopharma Investigational Site, Pavia
- Japan (21):
  - Theravance Biopharma Investigational Site, Nagoya, Aichi-ken
  - Theravance Biopharma Investigational Site, Abiko, Chiba
  - Theravance Biopharma Investigational Site, Sakura, Chiba
  - Theravance Biopharma Investigational Site, Kurume, Fukuoka
  - Theravance Biopharma Investigational Site, Ōgaki, Gifu
  - Theravance Biopharma Investigational Site, Isesaki, Gunma
  - Theravance Biopharma Investigational Site, Hatsukaichi, Hiroshima
  - Theravance Biopharma Investigational Site, Hiroshima, Hiroshima
  - Theravance Biopharma Investigational Site, Kawasaki, Kanagawa
  - Theravance Biopharma Investigational Site, Sendai, Miyagi
  - Theravance Biopharma Investigational Site, Suwa, Nagano
  - Theravance Biopharma Investigational Site, Ōita, Oita Prefecture
  - Theravance Biopharma Investigational Site, Fujiidera, Osaka
  - Theravance Biopharma Investigational Site, Izumiōtsu, Osaka
  - Theravance Biopharma Investigational Site, Ageo Shi, Saitama
  - Theravance Biopharma Investigational Site, Tokorozawa, Saitama
  - Theravance Biopharma Investigational Site, Kurobe-shi, Toyama
  - Theravance Biopharma Investigational Site, Chiba
  - Theravance Biopharma Investigational Site, Fukuoka
  - Theravance Biopharma Investigational Site, Kumamoto
  - Theravance Biopharma Investigational Site, Tokyo
- Poland (13):
  - Theravance Biopharma Investigational Site, Poznan, Greater Poland Voivodeship
  - Theravance Biopharma Investigational Site, Torun, Kuyavian-Pomeranian Voivodeship
  - Theravance Biopharma Investigational Site, Włocławek, Kuyavian-Pomeranian Voivodeship
  - Theravance Biopharma Investigational Site, Krakow, Lesser Poland Voivodeship
  - Theravance Biopharma Investigational Site, Wroclaw, Lower Silesian Voivodeship
  - Theravance Biopharma Investigational Site, Piaseczno, Masovian Voivodeship
  - Theravance Biopharma Investigational Site, Warsaw, Masovian Voivodeship
  - Theravance Biopharma Investigational Site, Sopot, Pomeranian Voivodeship
  - Theravance Biopharma Investigational Site, Tychy, Silesian Voivodeship
  - Theravance Biopharma Investigational Site, Szczecin, West Pomeranian Voivodeship
  - Theravance Biopharma Investigational Site, Świętokrzyskie
  - Theravance Biopharma Investigational Site, Ksawerów, Łódź Voivodeship
  - Theravance Biopharma Investigational Site, Lodz, Łódź Voivodeship
- Portugal (8):
  - Theravance Biopharma Investigational Site, Coimbra
  - Theravance Biopharma Investigational Site, Guimarães
  - Theravance Biopharma Investigational Site, Leiria
  - Theravance Biopharma Investigational Site, Lisbon
  - Theravance Biopharma Investigational Site, Santa Maria da Feira
  - Theravance Biopharma Investigational Site, Senhora da Hora
  - Theravance Biopharma Investigational Site, Viana do Castelo
  - Theravance Biopharma Investigational Site, Vila Nova de Gaia
- Romania (2):
  - Theravance Biopharma Investigational Site, Timișoara, Timiș County
  - Theravance Biopharma Investigational Site, Bucharest
- Serbia (5):
  - Theravance Biopharma Investigational Site, Belgrade
  - Theravance Biopharma Investigational Site, Kragujevac
  - Theravance Biopharma Investigational Site, Niš
  - Theravance Biopharma Investigational Site, Subotica
  - Theravance Biopharma Investigational Site, Zrenjanin
- Slovakia (3):
  - Theravance Biopharma Investigational Site, Prešov, Prešovsky
  - Theravance Biopharma Investigational Site, Nitra
  - Theravance Biopharma Investigational Site, Šahy
- Theravance Biopharma Investigational Site, Johannesburg, Gauteng, South Africa
- South Korea (4):
  - Theravance Biopharma Investigational Site, Wŏnju, Gangwon-do
  - Theravance Biopharma Investigational Site, Suwon, Gyeonggi-do
  - Theravance Biopharma Investigational Site, Daegu
  - Theravance Biopharma Investigational Site, Seoul
- Spain (4):
  - Theravance Biopharma Investigational Site, Barcelona
  - Theravance Biopharma Investigational Site, Madrid
  - Theravance Biopharma Investigational Site, Seville
  - Theravance Biopharma Investigational Site, Valencia
- Taiwan (4):
  - Theravance Biopharma Investigational Site, Kaohsiung City, Kaohsiung City
  - Theravance Biopharma Investigational Site, Taichung
  - Theravance Biopharma Investigational Site, Tainan
  - Theravance Biopharma Investigational Site, Taipei
- Ukraine (14):
  - Theravance Biopharma Investigational Site, Kiev, KIEV CITY
  - Theravance Biopharma Investigational Site, Kyiv, Kyiv City
  - Theravance Biopharma Investigational Site, Kremenchuk, Poltava Oblast
  - Theravance Biopharma Investigational Site, Uzhhorod, Transcarpathian
  - Theravance Biopharma Investigational Site #2, Vinnytsia, Vinnytsya
  - Theravance Biopharma Investigational Site, Vinnytsia, Vinnytsya
  - Theravance Biopharma Investigational Site, Uzhhorod, Zakarpattia Oblast
  - Theravance Biopharma Investigational Site, Chernivtsi
  - Theravance Biopharma Investigational Site, Kharkiv
  - Theravance Biopharma Investigational Site #2, Lviv
  - Theravance Biopharma Investigational Site, Lviv
  - Theravance Biopharma Investigational Site, Ternopil
  - Theravance Biopharma Investigational Site, Vinnytsia
  - Theravance Biopharma Investigational Site, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 46 out of the planned 500 participants were enrolled and received study drug between 23 July 2020 and 27 October 2021.
Groups:
- TD-1473 20mg: Participants received TD-1473 orally at a dose of 20mg once daily.
- TD-1473 80mg: Participants received TD-1473 orally at a dose of 80mg once daily.
- TD-1473 200mg: Participants received TD-1473 orally at a dose of 200mg once daily.
Period: Overall Study
Arm/Group | TD-1473 20mg | TD-1473 80mg | TD-1473 200mg
Started | 13 | 18 | 15
Completed | 0 | 0 | 0
Not Completed | 13 | 18 | 15
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 2
Not completed — Study Terminated By Sponsor | 12 | 17 | 12
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population includes all participants from the Safety Analysis Set. The Safety Analysis Set includes all participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | TD-1473 20mg | TD-1473 80mg | TD-1473 200mg | Total
Number analyzed (Participants) | 13 | 18 | 15 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.31 (17.375) | 43.22 (15.869) | 46.13 (13.432) | 45.04 (15.296)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 7 | 22
  Male | 5 | 11 | 8 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 12 | 17 | 15 | 44
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 3 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 12 | 15 | 13 | 40
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: A TEAE was defined as any AE with a recorded start date on or after the date of the first dose of study drug up through 4 weeks after the last dose of study drug. Any clinically significant changes in laboratory safety tests, electrocardiograms (ECGs) and vital signs, were also recorded as TEAEs.
Time Frame: Day 1 up to 4 weeks after last dose of study drug (median treatment duration was: TD-1473 20 mg - 142 days; TD-1473 80 mg - 180.0 days; TD-1473 200 mg - 158 days)
Population: Includes all participants from the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | TD-1473 20mg | TD-1473 80mg | TD-1473 200mg
Number analyzed (Participants) | 13 | 18 | 15
Participants | 4 | 5 | 6

ADVERSE EVENTS:
Time Frame: Day 1 up to 4 weeks after last dose of study drug (median treatment duration was: TD-1473 20 mg - 142 days; TD-1473 80 mg - 180.0 days; TD-1473 200 mg - 158 days)
Description: Includes all participants from the Safety Analysis Set.
Arm/Group | TD-1473 20mg | TD-1473 80mg | TD-1473 200mg
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/18 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/18 | 1/15
Other Adverse Events (participants affected / at risk) | 4/13 | 5/18 | 5/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TD-1473 20mg (N=13) | TD-1473 80mg (N=18) | TD-1473 200mg (N=15)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TD-1473 20mg (N=13) | TD-1473 80mg (N=18) | TD-1473 200mg (N=15)
COVID-19 (Infections and infestations) | 0 | 0 | 1
Chlamydial infection (Infections and infestations) | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Study 0164 was terminated early because Study 0157 was terminated early and participation in Study 0164 was predicated on participation in Study 0157.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT03920254/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/54/NCT03920254/SAP_001.pdf